CLINICAL TRIAL: NCT06232967
Title: Long-term Outcome of Primary Tumor Resection in Non-Small-Cell Lung Cancer Patients With Dry Pleural Dissemination: A Multi-center Study
Brief Title: PPIO-006 Primary Tumor Resection for IVa NSCLC
Status: Completed | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, WEI GUO, PhD., Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: Wei Guo
Record Dates: First submitted 2024-01-20; First posted 2024-01-31 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Non-small-cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nuclear Receptor Subfamily 4, Group A, Member 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary tumor resection (PTR group): includes wedge resection, segmentectomy, or lobectomy.
  Interventions: Procedure: Primary tumor resection or not
- Exploratory thoracotomy (ET group): JSimply open and close surgery.

INTERVENTIONS:
Procedure: Primary tumor resection or not — For patients with non-small-cell lung cancer (NSCLC) and dry pleural dissemination, surgical decisions to perform exploratory thoracotomy only or primary tumor resection with wedge resection, segmentectomy, or lobectomy were based on surgeon experience and patient preference.
  Groups: Primary tumor resection (PTR group)

SUMMARY:
The goal of this mutli-center observational study is toinvestigate the impact of primary tumor resection (PTR) on the long-term survival of patients with non-small-cell lung cancer (NSCLC) and dry pleural dissemination (DPD). The main question it aims to answer is: whether primary tumor resection improve long-term survival of NSCLC patients with dry pleural dissemination.

DETAILED DESCRIPTION:
Non-small-cell lung cancer (NSCLC) patients with dry pleural dissemination have poor survival rates and are generally contraindicated for surgery. Previous single-center retrospective studies have suggested that these patients may benefit from primary tumor resection (PTR). However, the evidence supporting PTR is still limited, especially in the era of targeted therapy. This study aimed to investigate the impact of PTR on the long-term survival of patients with NSCLC and DPD.

ELIGIBILITY:
Inclusion Criteria:

(1) pathologically confirmed primary NSCLC with malignant pleural dissemination, (2) no preoperative treatment, (3) age 80 years or younger, (4) clinicopathologic data and follow-up results were complete.

Exclusion Criteria:

(1) pleural effusion, contralateral lung metastasis or distant metastasis revealed preoperatively, and (2) with a history of other malignant disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2016 to December 2023, a total of 204 consecutive NSCLC patients with surgically confirmed DPD were collected retrospectively from three high-volume centers in China. Data were obtained by reviewing medical records.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Disease-specific survival (DSS) | Up to 8 years
  The duration from the day of surgery to the the last follow-up visit or to death specifically caused by NSCLC.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 8 years
  The duration of survival with no evidence of progression of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, PhD, Principal Investigator — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Army Medical Center of the People's Liberation Army, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bao T, Deng Y, Chen L, Sun W, Ge M, Zhao X, Chen X, Zhang L, Wang Y, He X, Pu X, He Y, Yu J, Guo W. Primary tumour resection in non-small cell lung cancer patients with pleural dissemination unexpectedly detected during operation: a two-centre retrospective cohort study. BMC Cancer. 2025 Feb 21;25(1):316. doi: 10.1186/s12885-025-13747-3. PMID 39984876